CLINICAL TRIAL: NCT02136628
Title: Posincisional Hernia Prevention. Effectiveness of Reinforced Tension Line (RTL) Technique Compared With the Conventional Method
Brief Title: Hernia Prevention. Effectiveness of Reinforced Tension Line (RTL) Technique Compared With the Conventional Method
Acronym: Herniapreven
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Jose Antonio de Jesus Alvarez Canales, Ph. D., Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-HRAEB_2013-020
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Hernia
Keywords: RTL Technique
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RTL (Experimental): The method consists of two lines of suture, each, over the fascial wound edge. It starts with a suture strand (in this study was used PDS number 0) in one end of the fascial wound where the suture is run longitudinally and parallel to the aponeurotic edge. The needle should go in and out at intervals of 1 cm away and always kept at 0.5 cm from the edge of the fascia. Upon reaching the opposite angle of the wound suture strand another repeating the same process on the fascial edge otherwise used. The ends of the two suture strands are tied in fascial angles.
  Thus the fascial wound is sutured with two lines of strengthening its edges. Then proceed to close the wound with continuous súrgete always ensuring that the suture lines remain anchored on suture reinforcement.
  Interventions: Procedure: Method RTL
- Control (No Intervention): Conventional midline mass closure technique. Upon completion of the surgical procedure was the closure of abdominal wall which will be made with the number 0 monofilament PDS, starting with knot at one end of the wound, continuous with continuous súrgete, moving each point to a centimeter away from the other. Each point will be a distance of one centimeter from the edge of the fascia. At the opposite end of the wound the same procedure was initiated and found the two suture lines at the midpoint of the wound will proceed to tying the two sutures with 4 square knots.

INTERVENTIONS:
Procedure: Method RTL — The method consists of two lines of suture, each, over the fascial wound edge. It starts with a suture strand (in this study was used PDS number 0) in one end of the fascial wound where the suture is run longitudinally and parallel to the aponeurotic edge. The needle should go in and out at intervals of 1 cm away and always kept at 0.5 cm from the edge of the fascia. Upon reaching the opposite angle of the wound suture strand another repeating the same process on the fascial edge otherwise used. The ends of the two suture strands are tied in fascial angles.
  Thus the fascial wound is sutured with two lines of strengthening its edges. Then proceed to close the wound with continuous súrgete always ensuring that the suture lines remain anchored on suture reinforcement.
  Arms: RTL

SUMMARY:
The posincisional hernia is considered a delicate complication , with an incidence of 10-12% in patients undergoing laparotomy may reach 45% in case of emergency and high-risk patients . It is estimated that in the United States are made about a million of reoperations for correction of this complication , with millions and despite the myriad studies that have been done in recent years there has been a decrease in the incidence losses and mortality of this complication.

Given the seriousness of this problem the last global consensus guidelines sent to the surgical community in three main areas: Identify the importance of the problem, improve the theoretical knowledge and technical capacity in the closure of the abdominal wall and Implement prophylaxis in selected patients.

The technique of reinforced tension line (RTL) was proposed by hollinsky and collaborators and is a strengthening of the abdominal incision with placement of a suture that runs lateral to the edge of the incision and closure of the abdominal wall is performed the usual manner with the only surgete continuous suture for closure is placed lateral to the suture reinforcement.

In the present study may contribute to these guidelines and to groups of patients at high risk were identified and applying the RTL technique and demonstrate that its use is safe and useful in reducing the presence of this complication could be implemented as prophylaxis handling the same .

The RTL method was applied experimentally on bodies to close the abdominal wall also be used in a cohort of patients for hernia repair wall , showing that by using it the abdominal wall is more resistant to shear forces by theoretical foundation that exists to show that could prevent the development of incisional hernias. There are no studies in the literature comparing this technique against conventional methods of closure of the abdominal wall as to the prevention of the same.

DETAILED DESCRIPTION:
The patient at the time of scheduled surgery either electively or urgently where planned preoperatively making approach by midline is invited to participate in the study, family and patient reported the details thereof and shall be obtained informed consent to participate.

The patient will be included in the experimental group (RTL) or (conventional) control according to a list of random numbers.

Estimated Enrollment: 76 Study Start Date July 2014 Estimated study completion date: May 2015 Estimated Primary Completion Date: January 2015.

Arms. Assigned interventions. Experimental: Procedure/ Surgery. Method RTL. The method consists of two lines of suture, each, over the fascial wound edge. It starts with a suture strand (in this study was used PDS number 0) in one end of the fascial wound where the suture is run longitudinally and parallel to the aponeurotic edge. The needle should go in and out at intervals of 1 cm away and always kept at 0.5 cm from the edge of the fascia. Upon reaching the opposite angle of the wound suture strand another repeating the same process on the fascial edge otherwise used. The ends of the two suture strands are tied in fascial angles.

Thus the fascial wound is sutured with two lines of strengthening its edges. Then proceed to close the wound with continuous súrgete always ensuring that the suture lines remain anchored on suture reinforcement.

Other Conventional midline mass closure technique. Upon completion of the surgical procedure was the closure of abdominal wall which will be made with the number 0 monofilament PDS, starting with knot at one end of the wound, continuous with continuous súrgete, moving each point to a centimeter away from the other. Each point will be a distance of one centimeter from the edge of the fascia. At the opposite end of the wound the same procedure was initiated and found the two suture lines at the midpoint of the wound will proceed to tying the two sutures with 4 square knots.

Participants surgeons evaluate the patient in the postoperative monitoring prior to hospital discharge , searching data hernia . After hospital discharge , participants surgeons evaluate the patient in the first external consultation with the attending surgeon looking data incisional hernia. Follow-up time will be 6 months which will be held in the outpatient and 6 months a CT will be made to identify the presence of incisional hernia

variables

Main outcome : presence of incisional hernia ( dichotomous categorical )

Secondary outcome : presence of complications of surgical wound ; infection , hematoma , ecchymosis , seroma ( categorical nominal)

Main predictor : technique for closure of the abdominal wall ( dichotomous categorical )

Conformation : gender ( dichotomous ) , age ( categorical nominal) , comorbidities ( categorical nominal) , emergency surgery ( dichotomous ), cough ( dichotomous ) , type of surgery ( categorical nominal) .

The presence of incisional hernia will be defined as loss of continuity of the abdominal wall after surgical closure , with the formation of a peritoneal sac and the protrusion of different structures of the cavity. Is clinically defined by the presence of a lump in the region of the surgical wound secondary to a physical effort as well as palpation of a defect in the continuity of the wound in the abdominal wall. The gold standard for diagnosis will be computed tomography in which the area of the disruption will be evaluated as well as the size and the organs involved , which will define the tomographic sign is the separation distance of the upright which should not be greater than 25 mm .

The present Study be made performed at the Hospital Regional de Alta Especialidad del Bajio.

Population. Patients over 18 years of age undergoing diagnostic laparotomy regardless of whether background urgent or scheduled at high risk for developing incisional hernia.

Universe:

Laparotomy patients scheduled for either elective or emergency with risk factors for developing incisional hernia.

Calculation of sample:

The sample size was calculated based on the study of Van Ramshorts, which found 40% of incisional hernia in patients at high risk with a score higher than 6 as the predictor scale, against 12% for the submission of the same in high-risk patients, earning a total of 76 patients, divided into 2 groups of 38 patients for each of the techniques, considering able to detect a difference of at least 28% in the proportion of patients without hernia, with 80% power and an alpha of 0.5% with two tails.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years undergoing elective or urgent laparotomy regardless of the underlying diagnosis .
* Patients who score 6 or higher on the scale of Van Ramshorst .
* Patients signed informed consent to participate in the study

Exclusion Criteria:

* Patients managed with open abdomen in those abdominal wall closure is not possible .
* Patients who do not have full data in the record and therefore are not classifiable according to the scale of Van Ramshorst .
* Patients for comorbidities and / or clinical status can not sign consent to participate in the study.
* Patients with history of previous midline laparotomy .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Posincisional hernia prevention | 6 months
  Participants surgeons evaluate the patient postoperatively until his discharge, and for 6 months in the outer query. the presence of incisional hernia will be determined in clinical fashion by the loss of continuity of the abdominal wall after surgical closure, with the formation of a peritoneal sac and the protrusion of different structures of the cavity, clinically by the presence of a bulge in the region of secondary wound a physical effort as well as palpation of a defect in the continuity of the wound in the abdominal wall. For diagnosis a CT scan in which the area of the disruption will be evaluated as well as the size and the organs involved, place the tomographic sign will define is the separation distance of the upright which must not exceed 25 mm.

REFERENCES:
- [Derived] Lozada-Hernandez EE, Mayagoitia-Gonzalez JC, Smolinski-Kurek RL, Montiel-Hinojosa L, Hernandez-Villegas L, Morales-Vargas JM, Perez-Sanchez KD, Orozco-Mosqueda A, Cano-Rosas M. Prevention of incisional hernia with a reinforced tension line (RTL) versus primary suture only in midline laparotomies: 3-year follow-up in a randomized clinical trial. Hernia. 2022 Apr;26(2):447-456. doi: 10.1007/s10029-020-02338-9. Epub 2021 Jan 5. PMID 33398464